CLINICAL TRIAL: NCT03843619
Title: Electronic and Lab Pre-screening of New Rheumatology Patients
Brief Title: Electronic and Lab Pre-screening of New Rheumatology Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Arthritis Northwest PLLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Discus Analytics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: R-17015
Record Dates: First submitted 2019-01-22; First posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Rheumatoid Arthritis; Inflammatory Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-E-referral: Patients who are referred in the traditional manner between two separate organizations.
- E-referral: Patients who are referred in an automated manner between two separate organizations.

SUMMARY:
By forming the foundation of a delivery system that integrates primary care (PC) and rheumatology, this initiative strives to strengthen the roles of both primary care and rheumatology practices as they co-manage patients in a quality care delivery system. Importantly, it strives to fill an unmet need, the rapid evaluation by Primary Care providers; the appropriate and timely referral of inflammatory disease patients to a rheumatologist; and the implementation of early aggressive therapy in the management of patients with rheumatoid arthritis (RA) with tight control. Given the call for improved quality, value, and demonstration of results[1], this initiative uses the tenets of National Center for Quality Assurance's Patient Centered Specialty Program[1] (PCSP) and it successfully masters and streamlines coordination of care.

ELIGIBILITY:
Inclusion Criteria:

* First ever referral to a rheumatologist.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to a rheumatologist for inflammatory arthritis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-02-28 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
To increase referral efficiencies through an electronic system to decrease the timeline prior | One year enrollment period
  Mean and median time (in days) to the first rheumatology visit from PCP referral for both cohorts

SECONDARY OUTCOMES:
To assess difference in disease activity progression using Clinical Disease Activity Index (CDAI) at both 12 and 24 months. | One year enrollment period with two year follow-up period.
  The change in CDAI score from baseline at 1 and 2 years. CDAI uses a scale of 0 - 60 where scores less than 2.8 are considered "remission", 2.9 - 10.0 are "low" disease activity, 10.1 - 22.0 are "moderate" disease activity, and 22.1 or higher are "high" disease activity.
To assess difference in disease activity progression using Routine Assessment of Patient Index Data (RAPID3) at both 12 and 24 months. | One year enrollment period with two year follow-up period.
  The change in RAPID3 score from baseline at 1 and 2 years. RAPID3 uses a scale of 0 - 30 where scores less than 3.1 are considered "remission", 3.1 - 6.0 are "low" disease activity, 6.1 - 12.0 are "moderate" disease activity, and 12.1 or higher are "high" disease activity.
To assess radiographic progression using sharp scores in the electronically referred cohorts versus the traditional cohort. | One year enrollment period with two year follow-up period.
  The change in sharp scores from baseline at 1 and 2 years.

IPD SHARING:
Plan to Share IPD: Undecided